CLINICAL TRIAL: NCT05251272
Title: A Combined Model Based on Spleen Stiffness, Liver Stiffness and Platelets for Assessing Portal Hypertension in Compensated Cirrhosis: A Prospective, Multicenter Study (CHESS2202)
Brief Title: A Combined Model Based on Spleen Stiffness, Liver Stiffness and Platelets for Assessing Portal Hypertension in Compensated Cirrhosis (CHESS2202)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: LanZhou University (Other); Shulan (Hangzhou) Hospital (Other); The Third People's Hospital of Taiyuan (Other); QuFu People's Hospital (Individual); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Prof., Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2202
Record Dates: First submitted 2022-01-28; First posted 2022-02-22 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Portal Hypertension
Keywords: compensated cirrhosis; spleen stiffness; liver stiffness; portal hypertension; hepatic venous pressure gradient
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Patients were fulfilled diagnosis of compensated cirrhosis based on radiological, histological features of liver cirrhosis and clinical manifestations.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient
- Validation cohort: Patients were fulfilled diagnosis of compensated cirrhosis based on radiological, histological features of liver cirrhosis and clinical manifestations.
  Interventions: Diagnostic Test: Hepatic venous pressure gradient

INTERVENTIONS:
Diagnostic Test: Hepatic venous pressure gradient — All patients underwent measurement of HVPG under local anesthesia.

SUMMARY:
Portal hypertension contributed to the main complications of liver cirrhosis. Currently, hepatic venous pressure gradient (HVPG) was the reference standard for evaluating portal pressure in patients with cirrhosis. However, the practice of HVPG is limited to require the extensive experience and highly specialized centers. In recent years, non-invasive methods were proposed to predict the degree of cirrhotic portal hypertension. Of them, liver stiffness measured by transient elastography had shown good performance for predicting clinically significant portal hypertension. However, liver stiffness only has a good correlation with portal pressure in the early stage of portal hypertension (HVPG<10 mmHg), because liver fibrosis is the main cause of portal hypertension in this period. In the stage of clinically significant portal hypertension (CSPH) (HVPG≥10 mmHg), increased portal vein inflow due to splanchnic vasodilation and hyperdynamic circulation, spleen stiffness may have a better correlation with HVPG than that of liver stiffness. Several studies have explored the combination of liver stiffness, platelet count and spleen stiffness for varices screening. However, there are few studies to report the above parameters for assessing CSPH and unneeded HVPG avoiding.

Since the spleen was stiffer than the liver, the current vibration-controlled transient elastography examination is dedicated to the liver, rather than the spleen. Very recently, a novel spleen-dedicated stiffness measured by transient elastography was proposed. The prospective, multicenter study aims to add spleen stiffness as a supplementary parameter to establish new criteria for identify CSPH in patients with compensated cirrhosis, with a dedicated probe on transient elastography equipment to assess spleen stiffness and liver stiffness, and further develop a novel model based on spleen stiffness for predicting the liver decompensation in patients with compensated cirrhosis.

DETAILED DESCRIPTION:
Portal hypertension contributed to the main complications of liver cirrhosis. Currently, hepatic venous pressure gradient (HVPG) was the reference standard for evaluating portal pressure in patients with cirrhosis. However, the practice of HVPG is limited to require the extensive experience and highly specialized centers. In recent years, non-invasive methods were proposed to predict the degree of cirrhotic portal hypertension. Of them, liver stiffness measured by transient elastography had shown good performance for predicting clinically significant portal hypertension. However, liver stiffness only has a good correlation with portal pressure in the early stage of portal hypertension (HVPG<10 mmHg), because liver fibrosis is the main cause of portal hypertension in this period. In the stage of clinically significant portal hypertension (CSPH) (HVPG≥10 mmHg), increased portal vein inflow due to splanchnic vasodilation and hyperdynamic circulation, spleen stiffness may have a better correlation with HVPG than that of liver stiffness. Several studies have explored the combination of liver stiffness, platelet count and spleen stiffness for varices screening. However, there are few studies to report the above parameters for assessing CSPH and unneeded HVPG avoiding.

Since the spleen was stiffer than the liver, the current vibration-controlled transient elastography examination is dedicated to the liver, rather than the spleen. Very recently, a novel spleen-dedicated stiffness measured by transient elastography was proposed. The prospective, multicenter study (leaded by The First Hospital of Lanzhou University and Shulan (Hangzhou) Hospital) aims to add spleen stiffness as a supplementary parameter to establish new criteria for identify CSPH in patients with compensated cirrhosis, with a dedicated probe on transient elastography equipment to assess spleen stiffness and liver stiffness, and further develop a novel model based on spleen stiffness for predicting the liver decompensation in patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. age above or equal to 18-year-old
2. fulfilled diagnosis of compensated cirrhosis based on radiological, histological features of liver cirrhosis and clinical manifestations
3. without decompensated events (e.g. ascites, bleeding, or overt encephalopathy)
4. with spleen stiffness and liver stiffness by a dedicated probe on transient elastography examination and platelet count measurement
5. with HVPG measurement
6. signed informed consent

Exclusion Criteria:

1. non-cirrhotic portal hypertension
2. accepted primary prevention (non-selective beta blockers or endoscopic variceal ligation)
3. lactation or pregnancy
4. suspicious or confirmed hepatocellular carcinoma
5. asplenia or splenectomy
6. incomplete clinical information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients was fulfilled the diagnosis of compensated cirrhosis based on radiological, histological features of liver cirrhosis and clinical manifestations.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Accuracy of a new model based on spleen stiffness (kPa), liver stiffness (kPa) or platelets (/L) for assessing portal hypertension in compensated cirrhosis. | 1 years
  In HVPG (mmHg) as reference method in evaluating portal pressure measured by intervention specialist, to develop a new model based on spleen stiffness (kPa), liver stiffness (kPa) or platelets (/L) and evaluate the accuracy in diagnosing portal hypertension.
  Spleen stiffness (kPa) and liver stiffness (kPa) are measured by transient elastography with a dedicated probe.

CONTACTS AND LOCATIONS:
Overall Officials: Lanjuan Li, M.D., Study Chair — Shulan (Hangzhou) Hospital; Xiaolong QI, M.D., Principal Investigator — LanZhou University; Huadong Yan, M.D., Study Director — Shulan (Hangzhou) Hospital
Locations (5):
- China (5):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Qufu People's Hospital, Jining, Shandong
  - The Third People's Hospital of Taiyuan, Taiyuan, Shanxi
  - Shulan (Hangzhou) Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Bureau C, Metivier S, Peron JM, Selves J, Robic MA, Gourraud PA, Rouquet O, Dupuis E, Alric L, Vinel JP. Transient elastography accurately predicts presence of significant portal hypertension in patients with chronic liver disease. Aliment Pharmacol Ther. 2008 Jun;27(12):1261-8. doi: 10.1111/j.1365-2036.2008.03701.x. Epub 2008 Apr 4. PMID 18397389
- [Background] Colecchia A, Montrone L, Scaioli E, Bacchi-Reggiani ML, Colli A, Casazza G, Schiumerini R, Turco L, Di Biase AR, Mazzella G, Marzi L, Arena U, Pinzani M, Festi D. Measurement of spleen stiffness to evaluate portal hypertension and the presence of esophageal varices in patients with HCV-related cirrhosis. Gastroenterology. 2012 Sep;143(3):646-654. doi: 10.1053/j.gastro.2012.05.035. Epub 2012 May 27. PMID 22643348
- [Background] Vizzutti F, Arena U, Romanelli RG, Rega L, Foschi M, Colagrande S, Petrarca A, Moscarella S, Belli G, Zignego AL, Marra F, Laffi G, Pinzani M. Liver stiffness measurement predicts severe portal hypertension in patients with HCV-related cirrhosis. Hepatology. 2007 May;45(5):1290-7. doi: 10.1002/hep.21665. PMID 17464971
- [Background] Colecchia A, Ravaioli F, Marasco G, Colli A, Dajti E, Di Biase AR, Bacchi Reggiani ML, Berzigotti A, Pinzani M, Festi D. A combined model based on spleen stiffness measurement and Baveno VI criteria to rule out high-risk varices in advanced chronic liver disease. J Hepatol. 2018 Aug;69(2):308-317. doi: 10.1016/j.jhep.2018.04.023. Epub 2018 May 3. PMID 29729368
- [Background] Pons M, Augustin S, Scheiner B, Guillaume M, Rosselli M, Rodrigues SG, Stefanescu H, Ma MM, Mandorfer M, Mergeay-Fabre M, Procopet B, Schwabl P, Ferlitsch A, Semmler G, Berzigotti A, Tsochatzis E, Bureau C, Reiberger T, Bosch J, Abraldes JG, Genesca J. Noninvasive Diagnosis of Portal Hypertension in Patients With Compensated Advanced Chronic Liver Disease. Am J Gastroenterol. 2021 Apr;116(4):723-732. doi: 10.14309/ajg.0000000000000994. PMID 33982942
- [Background] Stefanescu H, Marasco G, Cales P, Fraquelli M, Rosselli M, Ganne-Carrie N, de Ledinghen V, Ravaioli F, Colecchia A, Rusu C, Andreone P, Mazzella G, Festi D. A novel spleen-dedicated stiffness measurement by FibroScan(R) improves the screening of high-risk oesophageal varices. Liver Int. 2020 Jan;40(1):175-185. doi: 10.1111/liv.14228. Epub 2019 Sep 11. PMID 31444849
- [Background] Bastard C, Miette V, Cales P, Stefanescu H, Festi D, Sandrin L. A Novel FibroScan Examination Dedicated to Spleen Stiffness Measurement. Ultrasound Med Biol. 2018 Aug;44(8):1616-1626. doi: 10.1016/j.ultrasmedbio.2018.03.028. Epub 2018 May 3. PMID 29731186
- [Derived] Liu M, Zhang X, Cheng X, He Q, Zhou T, Wang H, Li B, Luo W, Li J, Li H, Lin Z, Song J, Wang W, Huang J, Ji Y, Zhou D, Xie W, Yang Q, Tu M, Luo X, Zhang X, Yan H, Chen J. Indocyanine Green Clearance Test via Pulse Dye Densitometry for Portal Hypertension Diagnosis in cACLD. Liver Int. 2025 Dec;45(12):e70425. doi: 10.1111/liv.70425. PMID 41178521